CLINICAL TRIAL: NCT06527560
Title: Clinical Trial Comparing Oral Versus Intravenous Cefuroxime in Pregnant Women with Pyelonephritis
Acronym: CEFURO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-0118
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pyelonephritis in Pregnancy
Keywords: pyelonephritis; pregnancy; cefuroxime
MeSH Terms: conditions — Pyelonephritis | interventions — Cefuroxime; cefuroxime axetil; Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: Randomized, parallel, non-inferiority trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients, care providers and investigators will not be aware of the treatment arm. Statistical analysis will be performed using pre-established criteria to access coded treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous cefuroxime (Active Comparator): Intravenous cefuroxime 750 mg every 8 hours + oral placebo every 12 hours
  Interventions: Drug: Cefuroxime
- Oral axetil cefuroxime (Experimental): Oral axetil cefuroxime 500 mg every 12 hours + intravenous saline solution every 8 hours
  Interventions: Drug: Cefuroxime Axetil

INTERVENTIONS:
Drug: Cefuroxime — Intravenous cefuroxime 750 mg every 8 hours
  Other Names: intravenous antibiotics + placebo Oral
  Arms: Intravenous cefuroxime
Drug: Cefuroxime Axetil — Oral cefuroxime 500 mg every 12 hours
  Other Names: oral antibiotics + placebo IV
  Arms: Oral axetil cefuroxime

SUMMARY:
The goal of this clinical trial is to compare rates of cure in pregnant women with pyelonephritis. The main question aims to answer:

Can we treat pyelonephritis in pregnancy with oral cefuroxime alone?

Pregnant women with pyelonephritis treated with intravenous cefuroxime will be the comparator.

Participants will be asked to accept participation in the study and will be randomly allocated to one of the two arms:

* Intravenous cefuroxime 750 mg every 8 hours + oral placebo every 12 hours
* Oral cefuroxime 500 mg every 12 hours + intravenous saline solution every 8 hours

DETAILED DESCRIPTION:
Urinary tract infections are common during pregnancy and can lead to pyelonephritis, a condition associated with morbidity in both the fetus and the pregnant woman. At HCPA, intravenous cefuroxime has been used until the antibiogram results from the pregnant woman's urine culture are available. However, this treatment requires hospitalization, which is financially burdensome and can affect the well-being of the pregnant woman. Despite this, there are not enough studies to investigate the use of oral cefuroxime as an initial treatment.

Objective: To compare the efficacy of cefuroxime administered orally versus intravenously in curing pyelonephritis during pregnancy, aiming to test the non-inferiority of the oral treatment.

Method: A randomized, prospective, triple-blind, two-arm study will be conducted. Pregnant women with pyelonephritis who agree to participate in the study at the time of hospitalization will receive the treatment: I) cefuroxime axetil 750mg IV every 8 hours and a placebo capsule 500mg; or II) 500mg orally every 12 hours and IV saline solution. These patients will be followed until the outcome is determined. After 48 hours in good clinical condition, the patients will be discharged and will continue treatment with cefuroxime axetil 500mg orally every 12 hours for 14 days. To analyze the difference in means and proportions with confidence intervals, Student's t-test will be performed, while nominal data will be analyzed using the chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 years or older and less than 20 weeks of gestational age, determined by ultrasound or the date of last menstruation, who come to the HCPA emergency department with a clinical diagnosis of pyelonephritis in pregnancy, defined as:
* Presence of lower back pain associated with
* Dysuria with leukocyturia, or hematuria or nitrite in the urine test with at least one of the criteria below:
* Leukocytosis (> 14,000 leukocytes/mL)
* Warm extremities, thready pulse, and tachycardia (HR > 110 bpm)
* Cyanosis and/or pallor
* Tachypnea (RR > 30 breaths/min)
* Arterial hypotension (SBP < 90mmHg)
* Positive costovertebral angle tenderness
* Urine culture with colony growth
* Hyperthermia (≥ 37.8°C)"

Exclusion Criteria:

* Do not wish to participate in the project.
* Used antimicrobials prior to hospitalization (3-day period).
* those who are allergic to cefuroxime.
* Have a urine culture antibiogram resistant to cefuroxime AND absence of clinical improvement (in this case, will be excluded as modified intention to treat).
* Have a diagnosis other than pyelonephritis, for example, appendicitis.
* those in septic shock, defined as:

  * the need for vasopressor to maintain a mean arterial pressure ≥ 65 mmHg and lactate > 2 mmol/l or 2 points on qSOFA. qSOFA will be considered positive when at least two of the following clinical criteria are present:
  * Respiratory rate greater than or equal to 22 breaths per minute;
  * Altered level of consciousness (Glasgow Coma Scale score less than 15);
  * Systolic blood pressure less than or equal to 100 mmHg.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnancy
Enrollment: 100 (Estimated)
Dates: Start 2024-09-09 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement | 3 days
  No fever, improvement of lower back pain
Negative urine culture | 21 days
  No growth of pathogenic bacteria in the urine culture

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo F Savaris, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- HCPA, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No
We did not decide what will be shared

REFERENCES:
- [Background] Ansaldi Y, Martinez de Tejada Weber B. Urinary tract infections in pregnancy. Clin Microbiol Infect. 2023 Oct;29(10):1249-1253. doi: 10.1016/j.cmi.2022.08.015. Epub 2022 Aug 27. PMID 36031053
- [Background] Blackwelder WC. "Proving the null hypothesis" in clinical trials. Control Clin Trials. 1982 Dec;3(4):345-53. doi: 10.1016/0197-2456(82)90024-1. PMID 7160191
- [Background] Faro S, Pastorek JG 2nd, Plauche WC, Korndorffer FA, Aldridge KE. Short-course parenteral antibiotic therapy for pyelonephritis in pregnancy. South Med J. 1984 Apr;77(4):455-7. doi: 10.1097/00007611-198404000-00011. PMID 6710201
- [Background] Finn A, Straughn A, Meyer M, Chubb J. Effect of dose and food on the bioavailability of cefuroxime axetil. Biopharm Drug Dispos. 1987 Nov-Dec;8(6):519-26. doi: 10.1002/bdd.2510080604. PMID 3427209
- [Background] Gilstrap LC 3rd, Cunningham FG, Whalley PJ. Acute pyelonephritis in pregnancy: an anterospective study. Obstet Gynecol. 1981 Apr;57(4):409-13. PMID 7243084
- [Background] Gilstrap LC 3rd, Ramin SM. Urinary tract infections during pregnancy. Obstet Gynecol Clin North Am. 2001 Sep;28(3):581-91. doi: 10.1016/s0889-8545(05)70219-9. PMID 11512502
- [Background] Powell N, Wade L, Iqbal-Elahi R, McDonald C, Philips R, Owens R, Amir A, Cho S, Nampa T, Lim D, Tai K, Jadav M. Potential impact of national recommendations to use short course antibiotic therapy on antibiotic use in the emergency department of a UK hospital: retrospective observational study. Eur J Hosp Pharm. 2022 Mar;29(2):72-78. doi: 10.1136/ejhpharm-2021-002756. Epub 2021 Nov 12. PMID 34772731
- [Background] Millar LK, Wing DA, Paul RH, Grimes DA. Outpatient treatment of pyelonephritis in pregnancy: a randomized controlled trial. Obstet Gynecol. 1995 Oct;86(4 Pt 1):560-4. doi: 10.1016/0029-7844(95)00244-l. PMID 7675380